CLINICAL TRIAL: NCT05190159
Title: Monster Screw System Post-Market Clinical Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Paragon 28 (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-SP-0001
Record Dates: First submitted 2021-12-20; First posted 2022-01-13 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Ankle Injuries; Foot Injury
MeSH Terms: conditions — Ankle Injuries; Foot Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Monster Screw System
  Interventions: Device: Monster Screw System

INTERVENTIONS:
Device: Monster Screw System — Subjects who have undergone a foot and/or ankle procedure involving the index device

SUMMARY:
Post-market clinical follow-up study on the Monster Screw System

DETAILED DESCRIPTION:
Ambispective, multi-surgeon, single site, consecutive case series to determine the safety, performance, and benefits of the Monster Screw System.

ELIGIBILITY:
Inclusion Criteria:

* The subject has undergone a foot and/or ankle procedure using the Monster Screw System and completed by one of the investigators.
* The subject has adequate radiographic and medical records

For the Prospective Data Collection:

- The subject is willing to provide written informed consent

Exclusion Criteria:

-None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigational population will include subjects who have undergone a foot and/or ankle procedure that fulfill the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Incidence of secondary procedures | Up to 9 months
  Safety will be assessed by recording the incidence of secondary procedures related to the index procedure
Incidence of adverse events | Up to 9 months
  Safety will be assessed by recording the incidence of adverse events

SECONDARY OUTCOMES:
Rate of Nonunion | Up to 9 months
  Safety as related to the rate of nonunion of the area treated with the index device
Rate of Maintenance of Correction | Up to 9 months
  Safety as related to the rate of the maintenance of correction
Rate of Index Device Failure | Up to 9 months
  Safety as related to the rate of the failure of the index device
Foot and Ankle Mobility Measure | Up to 54 months
  Device performance and benefits as related to Foot and Ankle Mobility Measure Activities of Daily Living (0-84) subscale and current level of daily activity rating (0-100). The higher the score, the higher the level of function, with 100% representing no dysfunction.
Visual Analog Scale | Up to 54 months
  Device performance and benefits as related to pain levels based on the Visual Analog Scale (range: 0 to 100; 0 = no pain; 100 = worst pain imaginable)
Patient satisfaction | Up to 54 months
  Device performance and benefits as related to patient satisfaction (very satisfied, good, fair, not satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jacy Legue, Study Director — Paragon 28
Locations (1):
- Henry Ford Health Systems, Jackson, Michigan, United States

IPD SHARING:
Plan to Share IPD: No